CLINICAL TRIAL: NCT04553068
Title: Phase 3 Double-blind Placebo-controlled Efficacy Trial of EVO100 Vaginal Gel for the Prevention of Urogenital Chlamydia Trachomatis and Neisseria Gonorrhoeae Infection
Brief Title: Evaluation of EVO100 for Prevention of Urogenital Chlamydia Trachomatis and Neisseria Gonorrhoeae Infection
Acronym: EVOGUARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EVO100-311
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sexually Transmitted Diseases; Gonorrhea; Chlamydia
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EVO100 gel (Experimental): EVO100 vaginal gel, 5 g
  Interventions: Drug: EVO100
- Placebo gel (Placebo Comparator): Placebo vaginal gel, 5 g
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EVO100 — EVO100 vaginal gel
  Arms: EVO100 gel
Drug: Placebo — Placebo vaginal gel
  Arms: Placebo gel

SUMMARY:
This study will evaluate whether EVO100 vaginal gel prevents the sexual transmission of CT and GC infection

DETAILED DESCRIPTION:
In this phase 3 double blind placebo controlled, efficacy study, women who have had a urogenital chlamydia or gonorrhea infection at any time over the 16 weeks preceding the enrollment Visit with one or more risk factors, or found to be positive for either infection at Screening Visit with one or more risk factors will be enrolled. After a screening period of up to 35 days, women will be randomized to receive either EVO100 vaginal gel or placebo. Each woman will participate in the study until she has completed 16 weeks of study medication or observation or tests positive for CT or GC infection.

ELIGIBILITY:
Subject Recruitment: EVOGUARDStudy.com/ct

Inclusion Criteria:

* Subjects must meet both of the following criteria:

  1. Urogenital CT and/or GC infection (documented in a retrievable medical record) within the 16 weeks prior to enrollment and one or more of the additional risk factors included below:

     * 18 to 24 years of age at the screening visit
     * New sex partner within the past 12 weeks (84 days)
     * More than one current sex partner
     * Knowledge that current sex partner has multiple partners
     * Partner with known sexually transmitted infection (STI)
     * Inconsistent condom use among persons who are not in a mutually monogamous relationship
  2. After three unsuccessful documented attempts to obtain medical records, the subject has a self-reported history of infection less than 17 weeks prior to enrollment AND two or more of the following additional risk factors:

     * 18 to 24 years of age at the screening visit
     * New sex partner within the past 12 weeks (84 days)
     * More than one current sex partner
     * Knowledge that current sex partner has multiple partners
     * Partner with known STI
     * Inconsistent condom use among persons who are not in a mutually monogamous relationship
* Ability to understand the consent process and procedures. For minors, the ability to obtain consent from parents/legal guardian and assent by minor subjects as applicable according to local regulations.
* Agree to be available for all study visits including Visit 5 and follow-up Visit 6 and comply with follow-up on staff appointment reminders
* Negative pregnancy test
* Negative CT and GC nucleic acid amplification test (NAAT) at screening or positive CT or GC NAAT and receives standard of care (SOC according to CDC or World Health Organization [WHO] guidelines) treatment prior to enrollment with subsequent negative CT and GC NAAT testing at enrollment visit
* Agree to use a woman-controlled method of contraception that is not directly delivered to the vaginal mucosa (with the exception of a vaginal ring) throughout the duration of the study, such as oral contraceptives, birth control implants, intrauterine devices (IUDs), or tubal ligation. Condom use only is not an acceptable form of contraception for this study
* Able and willing to comply with all study procedures, including the use of eDiaries and reporting of all Adverse Events and concomitant medications.
* Reports vaginal sexual intercourse with a male partner at least three times per month in the previous month and anticipates vaginal sexual intercourse regularly for the duration of the study
* Agree to abstain from douching or any form of vaginal suppository use (other than investigational product) during course of study

Exclusion Criteria:

* In the opinion of the Investigator, has a history of substance or alcohol abuse in the last 12 months or, has issues, conditions, or concerns that may compromise the safety of the subject, impact the subject's compliance with the protocol requirements, or confound the reliability of the data acquired
* Women who have undergone a total hysterectomy (had uterus and cervix removed). However, women with subtotal hysterectomy with an intact cervix may be enrolled
* Has a history or expectation of noncompliance with medications or intervention protocol
* Has engaged in sexual vaginal intercourse or douching, or used of any form of vaginal suppository or intravaginal device (with the exception of contraceptive vaginal ring or tampons) for 24 hours prior to enrollment (may be enrolled at a later date if all other criteria are met)
* Menstruating at enrollment (may be enrolled at a later date if all other criteria are met)
* Is currently being treated, or has been treated, for a period of 21 days prior to enrollment, with any prohibited antibiotics. The prohibited antibiotics include azithromycin, erythromycin, doxycycline, levofloxacin, ofloxacin, ceftriaxone, and cefixime.
* In the opinion of the Investigator, has signs/symptoms that indicate persistence of CT or GC infection diagnosed at screening, new interval infection, and/or a failure to comply with or complete the prescribed treatment regimen following a positive screening NAAT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females Only
Enrollment: 1892 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Maher, PhD, Study Director — Evofem Inc.
Locations (97):
- United States (97):
  - Cahaba Medical Care, Birmingham, Alabama
  - Mobile Obstetrics & Gynecology, P.C., Mobile, Alabama
  - Marchand OBGYN, Mesa, Arizona
  - Onyx Clinical Research, Peoria, Arizona
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Benchmark Research, Colton, California
  - Join Clinical Trials, Huntington Park, California
  - Matrix Clinical Research, Los Angeles, California
  - Dream Team Clinical Research, Pomona, California
  - Empire Clinical Research, Pomona, California
  - University of California, Davis Medical Center, Sacramento, California
  - UC San Diego Health, Womens Health Services La Jolla, San Diego, California
  - Providere Research Inc, West Covina, California
  - Planned Parenthood of Southern New England, New Haven, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Ideal Clinical Research, Aventura, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Homestead Associates in Research, Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Pharmax Research of South Florida, Inc, Miami, Florida
  - US Associates in Research, LLC, Miami, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Clintheory Healthcare Miami, North Miami Beach, Florida
  - Clinical Associates of Orlando, LLC, Orlando, Florida
  - Bioresearch Institute Llc, Pembroke Pines, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Comprehensive Clinical Research, LLC, West Palm Beach, Florida
  - Encore Medical Research of Weston, LLC, Weston, Florida
  - Visionaries Clinical Research, LLC, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Midtown OB GYN, Columbus, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Renew Health Clinical Research, Snellville, Georgia
  - University Women's Health Specialists, Honolulu, Hawaii
  - ASR,LLC, Nampa, Idaho
  - Eagle Clinical Research, Chicago, Illinois
  - Research Network America, Chicago, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Continental Clinical Solutions, Towson, Maryland
  - Boston Medical Center/Boston University Medical Campus, Boston, Massachusetts
  - Onyx Clinical Research, Flint, Michigan
  - Planned Parenthood North Central States - Minneapolis, Minneapolis, Minnesota
  - Lintecum and Nickell, P.C., Kansas City, Missouri
  - Planned Parenthood of the St. Louis Region and Southwest Missouri - Central West End Health Center, St Louis, Missouri
  - The Contraceptive Choice Center/Center for Outpatient Health - Women's Health Center, St Louis, Missouri
  - Planned Parenthood of Northern, Central and Southern New Jersey, Elizabeth, New Jersey
  - Planned Parenthood of Northern, Central and Southern New Jersey, Perth Amboy, New Jersey
  - Analyzed Health Clinical Trials, New York, New York
  - NYU Grossman School of Medicine/Bellevue Hospital Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Urgent Care Clinical Trials @ AFC Urgent Care-Bronx, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Circuit Clinical/OB GYN Associates of WNY, West Seneca, New York
  - Accellacare, Charlotte, North Carolina
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Across the LifeSpan, PLLC, Yanceyville, North Carolina
  - Seven Hills Clinical Research Group, Cincinnati, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Complete Healthcare For Women, Columbus, Ohio
  - DelRicht Research, Tulsa, Oklahoma
  - Planned Parenthood Columbia Willamette, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Planned Parenthood Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Magee-Womens Hospital, Center for Family Planning Research, Pittsburgh, Pennsylvania
  - Urgent Care Clinical Trials @ AFC Urgent Care-Easley, Easley, South Carolina
  - Urgent Care Clinical Trials @ AFC Urgent Care-Powdersville, Powdersville, South Carolina
  - Urgent Care Clinical Trials @ AFC Urgent Care-Clemson, Seneca, South Carolina
  - WR-Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - Urgent Care Clinical Trials @ Complete Health Care Partners, Nashville, Tennessee
  - Coastal Bend Clinical Research, Corpus Christi, Texas
  - Urgent Care Clinical Trials @City Doc Urgent Care - McKinney, Dallas, Texas
  - AIDS Arms, Inc. DBA Prism Health North Texas, Dallas, Texas
  - Urgent Care Clinical Trials @City Doc Urgent Care-Inwood, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - Synergy Groups Medical LLC, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Cypress Harmony Research, LLC, Houston, Texas
  - Encore Imaging and Medical Research, LLC, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Spring Family Practice Associates PA, Houston, Texas
  - MacArthur Medical Center, Irving, Texas
  - Maximos Ob/Gyn, League City, Texas
  - DCT-McAllen Primary Care Research dba Discovery Clinical Trials, McAllen, Texas
  - Centex Studies, Inc., McAllen, Texas
  - Synergy Groups Medical LLC, Missouri City, Texas
  - ARC Clinical Research at Kelly Lane, Pflugerville, Texas
  - Storks Research, LLC, Sugar Land, Texas
  - Virginia Women's Health Associates, Annandale, Virginia
  - TPMG Clinical Research, Newport News, Virginia
  - The Group for Women, Norfolk, Virginia
  - MultiCare Health System - Rockwood Clinic Cheney, Cheney, Washington
  - Planned Parenthood of the Great Northwest, Hawai'i, Alaska, Indiana, Kentucky - Tacoma Health Center, Tacoma, Washington

REFERENCES:
- [Derived] Thomas MA, Morlock R, Dart C, Howard B. Sexual Satisfaction Results With the Vaginal pH Modulator From the Phase 3 AMPOWER Study. J Sex Med. 2022 Jun;19(6):975-982. doi: 10.1016/j.jsxm.2022.03.221. Epub 2022 Apr 10. PMID 35418329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EVO100 Gel | Placebo Gel
Started | 943 | 949
Completed | 792 | 805
Not Completed | 151 | 144

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVO100 Gel | Placebo Gel | Total
Number analyzed (Participants) | 943 | 949 | 1892
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (10.31) | 29.7 (10.5) | 29.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 943 | 949 | 1892
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 467 | 447 | 914
  Not Hispanic or Latino | 461 | 482 | 943
  Unknown or Not Reported | 15 | 20 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 9 | 19
  Asian | 22 | 24 | 46
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 243 | 253 | 496
  White | 608 | 615 | 1223
  More than one race | 35 | 27 | 62
  Unknown or Not Reported | 23 | 19 | 42
Region of Enrollment [Number; unit: participants]
  United States | 943 | 949 | 1892

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Study Successes in the EVO100 and Placebo Treatment Groups
Description: Percentage of subjects who are defined study successes among the intervention groups with success defined as subjects completing the trial to Visit 5 without any CT or GC infection and no usage of prohibited antibiotics during the study.
Time Frame: 16 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 Gel | Placebo Gel
Number analyzed (Participants) | 906 | 913
Participants | 684 | 696

2. Secondary Outcome: Evaluate Safety of EVO100: AEs
Description: Descriptive analysis of AEs
Time Frame: 16 weeks
Population: Safety
Measure: Number; unit: participants
Arm/Group | EVO100 Gel | Placebo Gel
Number analyzed (Participants) | 926 | 937
participants
  Serious TEAEs | 4 | 9
  SAEs | 2 | 2
  Treatment related AEs | 81 | 62
  Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | EVO100 Gel | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/926 | 0/937
Serious Adverse Events (participants affected / at risk) | 4/926 | 9/937
Other Adverse Events (participants affected / at risk) | 39/926 | 28/937
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVO100 Gel (N=926) | Placebo Gel (N=937)
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
blood loss anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
alcohol poisoning (Nervous system disorders) | 1 (1) | 0 (0)
craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
fallopian tube abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tubo-ovarian abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pancreatic contusion (Hepatobiliary disorders) | 0 (0) | 1 (1)
abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVO100 Gel (N=926) | Placebo Gel (N=937)
vaginal discharge (Reproductive system and breast disorders) | 39 (39) | 28 (28) — vaginal discharge

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04553068/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04553068/SAP_001.pdf